CLINICAL TRIAL: NCT03548662
Title: The Effect of Platelet Rich Plasma Injection Combined With Exercise Rehabilitation in Patients With Rotator Cuff Tear
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-02-005B
Record Dates: First submitted 2017-10-10; First posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff Tear; Platelet Rich Plasma; Ultrasound; Exercise; Hyaluronic Acid
MeSH Terms: conditions — Rotator Cuff Injuries; Motor Activity | interventions — Hyaluronic Acid; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet-Rich Plasma Protein (PRP) Group (Experimental): Subjects in this group will receive PRP injection into tear site, followed by rehabilitative exercise
  Interventions: Biological: Platelet-Rich Plasma; Other: Exercise
- Hyaluronic Acid Group (Active Comparator): Subjects in this group will receive one injection with hyaluronic acid followed by rehabilitative exercise
  Interventions: Drug: Hyaluronic Acid; Other: Exercise

INTERVENTIONS:
Biological: Platelet-Rich Plasma — Platelet-Rich Plasma prepared by RegenKit® PRP, Regenlab SA
  Other Names: RegenKit® PRP
  Arms: Platelet-Rich Plasma Protein (PRP) Group
Drug: Hyaluronic Acid — Hyruan Plus Inj. produced by LG Life Sciences, Ltd.
  Other Names: Hyruan Plus Inj.
  Arms: Hyaluronic Acid Group
Other: Exercise — passive range of motion (PROM) exercise, active-assisted range of motion (AAROM) exercise, active range of motion (AROM) exercise, rotator cuff strengthening exercise, and peri-scapular muscle strengthening exercise

SUMMARY:
This study aims to evaluate the effect of platelet rich plasma combined with exercise therapy for patients with partial thickness rotator cuff tears.

DETAILED DESCRIPTION:
The purpose of this study is to exam the outcome of rotator cuff tear patients who received platelet rich plasma injection followed by rehabilitative exercise. The specific aim of this study is to determine the outcomes of treatment of partial thickness rotator cuff tears with platelet rich plasma (PRP) and rehabilitative exercise. Subjects with partial thickness rotator cuff tears will be designated to receive an injection of PRP or hyaluronic acid, followed by rehabilitative exercise. Shoulder function and tendon healing will be evaluated using the patient surveys as well as ultrasound. Subjects will be followed for 3 months to determine the outcomes of the treatment.

The hypothesis is that there is no difference in healing rate or functional outcomes in patients treated with PRP injections plus rehabilitative exercise compared with hyaluronic acid injection plus rehabilitative exercise for the treatment of partial thickness rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 85 years old, without significant cognition impairment (MMSE>20)
* Shoulder pain score(NRS)> 5
* Partial tear of supraspinatus tendon, proved by ultrasonography or MRI
* Patients who signed informed consent
* Patients who agreed to stop using analgesics during the experimental period

Exclusion Criteria:

* Thrombocytopenia (platelets less than 15000 per microliter)
* Patient who is using anticoagulant or has history of coagulation dysfunction
* Uncontrolled infection
* End stage malignant disease
* Infection or other skin condition over injection site
* History of shoulder or humeral fracture, dislocation or operation
* Psychiatric problems that precludes informed consent or inability to read or write
* Other serious problems that preclude participation of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Constant-Murley shoulder score | Change is measured from baseline to 1.5 and 3 months
  The Constant score assesses pain, function, ROM, and strength. Pain is allotted a maximum of 15 points, activities of daily living (function)20 points, ROM 40 points, and strength 25 points. The component scores are summated to achieve a maximum possible total score of 100.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Change is measured from baseline to 1.5 and 3 months
  The Numeric Pain Rating Scale (NRS) is a 11-point numeric scale ranges from '0' representing no pain to '10' representing worst pain imaginable
Shoulder range of motion | Change is measured from baseline to 1.5 and 3 months
  The shoulder range of motion (ROM) is measured in both active and passive manner and in four direction including flexion, extension, internal rotation and external rotation.
Shoulder Pain and Disability Index (SPADI) | Change is measured from baseline to 1.5 and 3 months
  SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. The scores from both domains are averaged to derive a total score with 0 being the best outcome (less disability) and 100 the worst (greater disability).
Size of rotator cuff tear | Change is measured from baseline to 1.5 and 3 months
  Rotator cuff tear size will be determined using ultrasound imaging. The image will be conducted in sagittal plan, transverse plan and will measure the maximal size of tear.

CONTACTS AND LOCATIONS:
Overall Officials: Jia chi Wang, MD, Principal Investigator — Taipei Veteran General hospital
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan